CLINICAL TRIAL: NCT02861768
Title: Improving the Diagnostic of Tuberculosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-49; 2012-A01598-35 (Registry Identifier: ansm)
Record Dates: First submitted 2016-08-05; First posted 2016-08-10 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2016-08

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- diagnosis of M.tuberculosis infection (Experimental)
  Interventions: Biological: Pharyngeal swab

INTERVENTIONS:
Biological: Pharyngeal swab

SUMMARY:
The presence of M. tuberculosis in non-invasive throat swabs of patients withdrawn for suspected tuberculosis.

Hypothesis 10% of patients infected by M. tuberculosis are carrier of M. tuberculosis pharyngeal.

Secondary

1. Measure the time to diagnosis of pulmonary TB by comparing the sample versus noninvasive pharyngeal samples taken routinely.
2. Evaluation of the direct cost of the diagnosis of M. tuberculosis by comparing the sample versus noninvasive pharyngeal samples taken routinely.
3. Beijing genotype prevalence among patients with pulmonary tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient taken for microbiological examinations "kit mycobacterium"
* Patient Major (> 18 years).
* Patient who freely signed the informed written consent.
* Patient affiliated to a system of social security. Exclusion criteria
* Patient minor (<18 years).
* Patient pregnant or nursing.
* Major Patient under guardianship.
* Private Patient liberty or under court order.
* Patient refusing to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 991 (Actual)
Dates: Start 2013-03-22; Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-08 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with microbiological diagnosis of M. tuberculosis infection | 3 years

SECONDARY OUTCOMES:
pulmonary tuberculosis diagnostic time. | 3years
Prevalence of diagnosed patients Beijing | 3 years
Direct cost of microbiological diagnosis of extra Beijing genotype | 3 years
  (compared to the cost of the kit TB), reported the percentage of patients diagnosed Beijing.

CONTACTS AND LOCATIONS:
Overall Officials: catherine GEINDRE, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France